CLINICAL TRIAL: NCT02516540
Title: Prospective Randomized Multicenter Trial to Assess the Efficacy of a Structured Physical Exercise Training and Mediterranean Diet in Women With BRCA1/2 Mutations
Brief Title: Efficacy of Lifestyle Intervention in BRCA1/2 Mutation Carriers
Acronym: LIBRE-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: University of Hohenheim (Other); University Hospital Schleswig-Holstein (Other); University of Leipzig (Other); University of Cologne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LIBRE-2-20150626
Record Dates: First submitted 2015-07-22; First posted 2015-08-06 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Hereditary Breast and Ovarian Cancer
Keywords: hereditary breast and ovarian cancer (HBOC); BRCA1/2 mutation carriers; Mediterranean diet; Structured exercise training; prevention
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Study participants are instructed regarding a healthy diet according to the recommendations of the German Nutrition Society (DGE) and are informed about positive effects of physical activity on incidence and prognosis of breast cancer
- Intervention (Experimental): Structured exercise training plus mediterranean diet: Study participants receive a lifestyle intervention of 12 months duration (3 months intensive intervention plus 9 months maintenance using monthly contacts and meetings). The intervention comprises a structured intensified training based on the results of physical performance diagnostics and a nutrition program based on a mediterranean diet.
  Interventions: Behavioral: Structured exercise training plus mediterranean diet

INTERVENTIONS:
Behavioral: Structured exercise training plus mediterranean diet — Structured exercise training plus mediterranean diet
  Arms: Intervention

SUMMARY:
The hypothesis of this 3 year, prospective randomized multicenter efficacy trial is that a structured life-style intervention program with exercise training and mediterranean diet is effective regarding increased adherence to a mediterranean diet, reduction of body mass index, and increase of physical fitness.

DETAILED DESCRIPTION:
BRCA1/2 mutation carriers have a considerably increased risk to develop breast and ovarian cancer during their lifetime. There is evidence from the literature that for sporadic breast cancer disease risk and the course of disease can be significantly influenced by physical activity, nutrition and weight. The hypothesis of this 3 year, prospective randomized multicenter efficacy trial is that a structured life-style intervention program with exercise training and mediterranean diet is effective regarding increased adherence to a mediterranean diet, reduction of body mass index, and increase of physical fitness.

ELIGIBILITY:
Inclusion Criteria:

* proven pathogenic BRCA1/2 mutation
* age >=18
* written informed consent

Exclusion Criteria:

* current chemotherapy of radiotherapy (inclusion 6 weeks after CTX or RX possible)
* metastatic tumor disease
* life expectancy <3 years
* clinically limiting cardiovascular or respiratory disease (instable CVD, heart failure stage IV, COPD GOLD IV, maximum resting blood pressure 160/100 mmHg)
* significant orthopedic disability which prevents from participating in the group interventions
* severe concomitant diseases which prevents from participating in the group interventions
* Karnofsky index <60
* maximum exercise capacity <50 W
* food allergies which prevent from mediterranean diet
* vegan diet
* body mass index <15 kg/m2
* pregnancy
* insufficient knowledge of German language
* insufficient compliance
* active participation in other interventional trials

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Mediterranean Diet Adherence Screener (MEDAS) Score (Questionnaire) | 12 months
  Adherence to mediterranean diet
body mass index (BMI) | 12 months
  Body weight (in kilograms) divided by body height (in meters) squared.
ventilatory threshold 1 (VT1) in spiroergometry | 12 months
  ventilatory threshold VT1 in spiroergometry

SECONDARY OUTCOMES:
stress coping capacity, as measured by the Trier Inventory for Chronic Stress (TICS) questionnaire | 3, 12, 24, 36 months
  (TICS) questionnaire
grade of optimism, as measured by the Life Orientation Test (LOT) questionnaire | 3, 12, 24, 36 months
  Life Orientation Test (LOT)
attitudes and beliefs regarding physical training and healthy diet, as measured by the "Bewertung körperlicher Aktivität und Ernährung" (BKAE) questionnaire | 3, 12, 24, 36 months
  (BKAE) questionnaire
quality of life, as measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | 3, 12, 24, 36 months
  (EORTC QLQ-C30)
maximum oxygen consumption (VO2max), as measured by spiroergometry | 3, 12 months
  spiroergometry
physical activity, as measured by the International Physical Activity Questionnaire (IPAQ) | 3, 12, 24, 36 months
  Physical Activity
incidence of breast cancer | 12, 24, 36 months
  During study
Mediterranean Diet Adherence Screener (MEDAS) Score | 3, 6, 9, 12, 24, 36 months
  (MEDAS) Score
body mass index (BMI) | 3, 12, 24, 36 months
  (BMI)
change of maximum oxygen consumption (VO2max) at ventilation threshold 1 (VT1), as measured by spiroergometry | 3, 12 months
  spiroergometry
mortality rate | 12, 24, 36 months
  During study
satisfaction (questionnaire) | 3, 12, 24, 36 months
  satisfaction (questionnaire)
tobacco consumption | 12, 24, 36 months
  survey
alcohol consumption | 12, 24, 36 months
  survey
dietary habits and calory intake, as measured by the European Prospective Investigation into Cancer and Nutrition Study Food Frequency Questionnaire (EPIC-FFQ) | 3, 12, 24, 36 months
  (EPIC-FFQ)
serum cholesterol, serum high density lipoprotein cholesterol,serum, serum Glucose, triglycerides, c-reactive Protein, serum Insulin,proneurotensin | 3, 12, 24, 36 months
  Blood Test
proenkephalin | 3, 12, 24, 36 months
  Genetic test
Omega 3 fatty acid in the erythrocyte Membrane, Omega 6 fatty acid level in the erythrocyte Membraserum low density, lipoprotein cholesterolne, Omega 9 fatty acid level in the erythrocyte Membrane, | 3, 12, 24, 36 months
  Blood Test

CONTACTS AND LOCATIONS:
Overall Officials: Marion Kiechle, Prof. Dr., Study Director — Technical University of Munich; Martin Halle, Prof. Dr., Study Director — Technical University of Munich; Stephan C Bischoff, Prof. Dr., Study Director — Universitaet Hohenheim, Stuttgart; Michael Siniatchkin, Prof. Dr., Study Director — University Hospital Schleswig-Holstein; Markus Loeffler, Prof. Dr., Study Director — University of Leipzig; Christoph Engel, PD Dr., Study Director — University of Leipzig; Rita K Schmutzler, Prof. Dr., Study Director — University of Cologne; Alfons Meindl, Prof. Dr., Study Director — Technical University of Munich; Anne S Quante, Dr., Principal Investigator — Technical University of Munich
Locations (19):
- Germany (19):
  - Humboldt Universität zu Berlin, Berlin
  - Uniklinikum Köln, Cologne
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Kliniken Essen-Mitte, Essen
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinium Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Technische Universität München, München
  - Universität Regensburg, Regensburg
  - Interdisziplinäres Brustzentrum am Diakonieklinikum, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
  - Universität Ulm, Ulm
  - Universitätsklinikum Würzburg, Würzburg

REFERENCES:
- [Derived] Seethaler B, Nguyen NK, Basrai M, Kiechle M, Walter J, Delzenne NM, Bischoff SC. Short-chain fatty acids are key mediators of the favorable effects of the Mediterranean diet on intestinal barrier integrity: data from the randomized controlled LIBRE trial. Am J Clin Nutr. 2022 Oct 6;116(4):928-942. doi: 10.1093/ajcn/nqac175. PMID 36055959
- [Derived] Kiechle M, Engel C, Berling A, Hebestreit K, Bischoff SC, Dukatz R, Siniatchkin M, Pfeifer K, Grill S, Yahiaoui-Doktor M, Kirsch E, Niederberger U, Enders U, Loffler M, Meindl A, Rhiem K, Schmutzler R, Erickson N, Halle M. Effects of lifestyle intervention in BRCA1/2 mutation carriers on nutrition, BMI, and physical fitness (LIBRE study): study protocol for a randomized controlled trial. Trials. 2016 Jul 29;17:368. doi: 10.1186/s13063-016-1504-0. PMID 27473440